CLINICAL TRIAL: NCT02452424
Title: Phase 1/2a Study of Double-Immune Suppression Blockade By Combining a CSF1R Inhibitor (PLX3397) With An Anti-PD-1 Antibody (Pembrolizumab) To Treat Advanced Melanoma And Other Solid Tumors
Brief Title: A Combination Clinical Study of PLX3397 and Pembrolizumab To Treat Advanced Melanoma and Other Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated early for insufficient evidence of clinical efficacy
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Plexxikon (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLX108-14; KEYNOTE-103 (Other: Merck Sharp & Dohme Corp.)
Record Dates: First submitted 2015-05-20; First posted 2015-05-22 (Estimated); Results first posted 2019-10-09 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-02

CONDITIONS: Melanoma; Non-small Cell Lung Cancer; Squamous Cell Carcinoma of the Head and Neck; Gastrointestinal Stromal Tumor (GIST); Ovarian Cancer
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Gastrointestinal Stromal Tumors; Ovarian Neoplasms | interventions — pexidartinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PLX3397 and Pembrolizumab (Part 1) (Experimental): Open-label, sequential PLX3397 dose escalation with a fixed dose of pembrolizumab in approximately 24 patients with advanced solid tumors.
  (Enrollment complete- 33 enrolled)
  Interventions: Drug: PLX3397; Biological: Pembrolizumab
- PLX3397 and Pembrolizumab (Part 2) (Experimental): Extension cohort at the RP2D of PLX3397 in combination with pembrolizumab in approximately 376 patients with advanced solid tumors
  (Enrollment Complete- 45 enrolled)
  Interventions: Drug: PLX3397; Biological: Pembrolizumab

INTERVENTIONS:
Drug: PLX3397 — PLX3397 capsules, 200 mg
  Other Names: Pexidartinib
Biological: Pembrolizumab — Pembrolizumab, 200 mg, IV
  Other Names: Keytruda, MK-3475, SCH 900475

SUMMARY:
The goal of this clinical research study is to learn how PLX3397 and pembrolizumab work together to affect cancer cells.

PLX3397 is designed to target the receptor for CSF1 (CSF1R). Pembrolizumab is designed to block the interaction between the receptor PD-1 and molecules that bind PD-1. In this study, PLX3397 and pembrolizumab are being given together in order to study their combined effects on patients' immune responses to their tumors. Tumor-specific immune responses have been shown to kill cancer cells and/or to stop tumors from growing.

Part 1 of the study (dose-escalation phase) will establish the safest dose of PLX3397 to be given in combination with pembrolizumab. Part 2 of the study (expansion phase) will include an evaluation of efficacy of this combination in the following tumor types:

* Advanced melanoma: prior anti-PD-1/PD-L1 therapy but never responded
* Advanced melanoma: prior anti-PD-1/PD-L1 therapy and responded but later progressed as defined by irRECIST while on therapy
* Non-small cell lung cancer
* Ovarian cancer
* Gastrointestinal Stromal Tumor (GIST)
* Squamous cell cancer of the head and neck

ELIGIBILITY:
Inclusion Criteria:

A subject must satisfy all of the following criteria to be considered for inclusion in the study:

* Subjects with histologically or cytologically-confirmed diagnosis of cancer that is recurrent, metastatic, or persistent, who have relapsed from or are refractory to treatment and who also meet the following corresponding requirements for the cohort or phase of the study into which they will enroll:
* Dose-escalation Phase: Subjects with advanced solid tumors (any tumor type) considered to have no standard-of care treatment for their malignancy with a curative intent, either as initial therapy or after progressing to prior therapies; subjects who have been treated previously with a CSF1R inhibitor or an anti PD1/PDL1 inhibitor may enroll.
* Expansion Phase: Subjects with 1 of the tumor types who have relapsed from or are refractory to standard treatment. Subjects with non-small-cell lung cancer (non-squamous; EGFR, ALK wild type), advanced melanoma, ovarian cancer, unresectable RCC with component of clear-cell histology and/or component of sarcomatoid histology, glioblastoma or gliosarcoma, gastrointestinal stromal tumor.
* Subjects with melanoma must have a histologically confirmed diagnosis of stage III disease not amenable to local therapy. Melanoma subjects may have received any number of prior lines of therapy for metastatic disease and must have measurable disease per RECISTv1.1. Subjects with melanoma who have received prior treatment with a BRAF/MEK inhibitor are acceptable candidates.
* Expansion cohorts: Subjects must have relapsed or been refractory to standard treatment. NSCLC, SCCHN, and Melanoma must show primary progression with antiPD1/anti-PDL1 therapy. They must have tumor accessible for sequential biopsy (core needle biopsy or excision required) and be willing to provide on study tumor tissue biopsy. Subjects for whom newly obtained samples cannot be obtained (e.g. inaccessible or patient safety concern) may submit an archived specimen onlyupon agreement from the Sponsor.
* ECOG performance status 0 or 1.
* Women of childbearing potential must have a negative serum pregnancy test within 72 hours prior to initiation of dosing.
* Women of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Women of non-child bearing potential may be included if they are either surgically sterile or have been postmenopausal for ≥1 year.
* Fertile men must agree to use an effective method of birth control starting with the first dose of study treatment through 120 days after the last dose of study treatment.
* Adequate organ function as demonstrated by laboratory values.

Exclusion Criteria:

A subject who meets any of the following criteria will be disqualified from entering the study:

* Disease that is suitable for local therapy administered with curative intent.
* Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment.
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 28 days prior to the first dose of study treatment.
* Has had monoclonal antibody within 28 days of first dose of study treatment or has not recovered from AEs due to agents administered more than 28 days earlier.
* Has had chemotherapy, targeted small molecule therapy, or radiation therapy within 14 days prior to first dose of study treatment or who has not recovered from AEs due to a previously administered agent.
* Note: Subjects with ≤ Grade 2 neuropathy or ≤ Grade 2 alopecia are an exception to this criterion and may qualify for the study.
* Note: If a subject received major surgery, he or she must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
* Has received transfusion of blood products (including platelets or red blood cells [RBC]) or administration of colony stimulating factors (including granulocyte colony-stimulating factor, granulocyte macrophage colony-stimulating factor, or recombinant erythropoietin) within 28 days prior to Day 1.
* Evidence of interstitial lung disease or active, noninfectious pneumonitis.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy, in situ cervical cancer and isolated elevation of prostate-specific antigen. Subjects with a completely treated prior malignancy with no evidence of disease for ≥ 2 years are eligible.
* For Dose escalation cohort: patients with liver metastases, inclusion of patients with liver metastases in subsequent cohorts will be based upon clinical data.
* For Expansion cohort subjects who have previously received an anti-PD-1, anti-PD-L1, or anti#PD-L2 agent or has previously participated in pembrolizumab clinical trials are excluded, except the following tumor types Melanoma, NSCLC and SCCHN (who must show primary progression to anti-PD1/anti-PDL1 therapy).
* Radiation therapy within 14 days of first dose of study treatment.- remove since it's repetitive
* Has active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy is not considered a form of systemic treatment.
* Has an active infection requiring systemic therapy.
* Has known central nervous system metastases and/or carcinomatous meningitis.

  o Note: Subjects with previously treated brain metastases may participate if they meet the following criteria: 1) are stable for at least 28 days prior to the first dose of study treatment and if all neurologic symptoms returned to baseline); 2) have no evidence of new or enlarging brain metastases; and 3) have not been using steroids for at least 7 days prior to first dose of study treatment. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability.
* Uncontrolled intercurrent illness.
* Refractory nausea and vomiting, malabsorption, external biliary shunt, or significant small bowel resection that would preclude adequate absorption.
* QT interval corrected using Fridericia's formula (QTc) ≥ 450 msec (males) or ≥ 470 msec (females) at Screening.
* Congenital long QT syndrome or patients taking concomitant medications known to prolong the QT interval.
* Major surgery within 28 days prior to first dose of study treatment.
* Has received a live vaccine administered within 30 days prior to first dose of study treatment.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Active and clinically significant bacterial, fungal or viral infection, including hepatitis B virus (HBV), hepatitis C virus (HCV), known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome related illness (HIV testing is not required), including subjects who have an active infection requiring systemic therapy.
* Any of the following within 48 weeks (~1 year) prior to first dose of study treatment: myocardial infarction, uncontrolled angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of study treatment.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Has had prior exposure to PLX3397.
* Has had hypersensitivity (≥Grade 3) reaction to pembrolizumab and/or any of its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2015-07-02 (Actual); Primary Completion 2018-08-17 (Actual); Study Completion 2018-10-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Marin Cancer Care, Greenbrae, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University St. Louis Siteman Cancer Center, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Medical University Health Hollings Cancer Center, Charleston, South Carolina
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https:// vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dose Escalation: 33 participants who met the inclusion and none of the exclusion criteria were enrolled and received study drug.
  Dose Expansion: 45 participants with melanoma, non-small cell lung cancer (NSCLC), ovarian cancer, squamous cell carcinoma of the head and neck (SCCHN), and gastrointestinal stromal tumor (GIST) were enrolled.
Pre-assignment Details: Dose Escalation: Up to 42 participants with advanced solid tumors (any type) were to be enrolled sequentially in up to 7 cohorts (3+3 design).
  Dose Expansion: Up to 483 participants were planned with the sample size for each tumor type based on a truncated sequential probability ratio test (max sample size 28 to 48 participants per tumor type).
Groups:
- Dose Escalation: 400 mg/Day: Participants received pembrolizumab 200 mg IV every 3 weeks in combination with PLX3397 at 400 mg/day (administered twice daily [BID] as a split dose of 200 mg in the morning and 200 mg in the evening).
- Dose Escalation: 600 mg/Day: Participants received pembrolizumab 200 mg IV every 3 weeks in combination with PLX3397 at 600 mg/day (administered twice daily [BID] as a split dose of 200 mg in the morning and 400 mg in the evening).
- Dose Escalation: 600 mg/Day (Liver Metastases: Participants with liver metastases received pembrolizumab 200 mg IV every 3 weeks in combination with PLX3397 at 600 mg/day (administered twice daily [BID] as a split dose of 200 mg in the morning and 400 mg in the evening).
- Dose Escalation: 600 mg/Day (no Liver Metastases): Participants with no liver metastases received pembrolizumab 200 mg IV every 3 weeks in combination with PLX3397 at 600 mg/day (administered twice daily [BID] as a split dose of 200 mg in the morning and 400 mg in the evening).
- Dose Escalation: 800 mg/Day (Liver Metastases): Participants with liver metastases received pembrolizumab 200 mg IV every 3 weeks in combination with PLX3397 at 800 mg/day (administered twice daily [BID] as a split dose of 400 mg in the morning and 400 mg in the evening).
- Dose Escalation: 800 mg/Day (no Liver Metastases): Participants with no liver metastases received pembrolizumab 200 mg IV every 3 weeks in combination with PLX3397 at 800 mg/day (administered twice daily [BID] as a split dose of 400 mg in the morning and 400 mg in the evening).
- Dose Expansion: Melanoma: Participants with melanoma received pembrolizumab 200 mg IV every 3 weeks in combination with PLX3397 at 600 mg/day (administered twice daily [BID] as a split dose of 200 mg in the morning and 400 mg in the evening).
- Dose Expansion: NSCLC: Participants with NSCLC received pembrolizumab 200 mg IV every 3 weeks in combination with PLX3397 at 600 mg/day (administered twice daily [BID] as a split dose of 200 mg in the morning and 400 mg in the evening).
- Dose Expansion: Ovarian Cancer: Participants with ovarian cancer received pembrolizumab 200 mg IV every 3 weeks in combination with PLX3397 at 600 mg/day (administered twice daily [BID] as a split dose of 200 mg in the morning and 400 mg in the evening).
- Dose Expansion: SCCHN: Participants with SCCHN received pembrolizumab 200 mg IV every 3 weeks in combination with PLX3397 at 600 mg/day (administered twice daily [BID] as a split dose of 200 mg in the morning and 400 mg in the evening).
- Dose Expansion: GIST: Participants with GIST received pembrolizumab 200 mg IV every 3 weeks in combination with PLX3397 at 600 mg/day (administered twice daily [BID] as a split dose of 200 mg in the morning and 400 mg in the evening).
Period: Overall Study
Arm/Group | Dose Escalation: 400 mg/Day | Dose Escalation: 600 mg/Day | Dose Escalation: 600 mg/Day (Liver Metastases | Dose Escalation: 600 mg/Day (no Liver Metastases) | Dose Escalation: 800 mg/Day (Liver Metastases) | Dose Escalation: 800 mg/Day (no Liver Metastases) | Dose Expansion: Melanoma | Dose Expansion: NSCLC | Dose Expansion: Ovarian Cancer | Dose Expansion: SCCHN | Dose Expansion: GIST
Started | 4 | 3 | 7 | 9 | 4 | 6 | 13 | 8 | 15 | 3 | 6
Completed | 2 | 0 | 0 | 1 | 2 | 5 | 3 | 4 | 9 | 1 | 4
Not Completed | 2 | 3 | 7 | 8 | 2 | 1 | 10 | 4 | 6 | 2 | 2
Not completed — Death | 2 | 2 | 2 | 6 | 2 | 0 | 5 | 1 | 3 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Not completed — Other | 0 | 0 | 1 | 0 | 0 | 1 | 4 | 3 | 0 | 0 | 1
Not completed — Progressive disease (per RECIST) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Dose Escalation: 400 mg/Day: Participants received pembrolizumab 200 mg IV every 3 weeks in combination with of PLX3397 at 400 mg/day (administered twice daily [BID] as a split dose of 200 mg in the morning and 200 mg in the evening)..
- Dose Escalation: 600 mg/Day: Participants received pembrolizumab 200 mg IV every 3 weeks in combination with of PLX3397 at 600 mg/day (administered twice daily [BID] as a split dose of 200 mg in the morning and 400 mg in the evening).
- Dose Escalation: 600 mg/Day (Liver Metastases: Participants with liver metastases received pembrolizumab 200 mg IV every 3 weeks in combination with of PLX3397 at 600 mg/day (administered twice daily [BID] as a split dose of 200 mg in the morning and 400 mg in the evening).
- Dose Escalation: 600 mg/Day (no Liver Metastases): Participants with no liver metastases received pembrolizumab 200 mg IV every 3 weeks in combination with of PLX3397 at 600 mg/day (administered twice daily [BID] as a split dose of 200 mg in the morning and 400 mg in the evening).
- Dose Escalation: 800 mg/Day (Liver Metastases): Participants with liver metastases received pembrolizumab 200 mg IV every 3 weeks in combination with of PLX3397 at 800 mg/day (administered twice daily [BID] as a split dose of 400 mg in the morning and 400 mg in the evening).
- Dose Escalation: 800 mg/Day (no Liver Metastases): Participants with no liver metastases received pembrolizumab 200 mg IV every 3 weeks in combination with of PLX3397 at 800 mg/day (administered twice daily [BID] as a split dose of 400 mg in the morning and 400 mg in the evening)..
- Total: Total of all reporting groups
Arm/Group | Dose Escalation: 400 mg/Day | Dose Escalation: 600 mg/Day | Dose Escalation: 600 mg/Day (Liver Metastases | Dose Escalation: 600 mg/Day (no Liver Metastases) | Dose Escalation: 800 mg/Day (Liver Metastases) | Dose Escalation: 800 mg/Day (no Liver Metastases) | Dose Expansion: Melanoma | Dose Expansion: NSCLC | Dose Expansion: Ovarian Cancer | Dose Expansion: SCCHN | Dose Expansion: GIST | Total
Number analyzed (Participants) | 4 | 3 | 7 | 9 | 4 | 6 | 13 | 8 | 15 | 3 | 6 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 6 | 7 | 0 | 3 | 9 | 6 | 10 | 2 | 4 | 50
  >=65 years | 3 | 1 | 1 | 2 | 4 | 3 | 4 | 2 | 5 | 1 | 2 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (8.6) | 54.7 (10.2) | 51.1 (17.0) | 55.9 (10.9) | 72.0 (5.3) | 61.7 (8.7) | 61.8 (8.3) | 57.0 (11.3) | 60.4 (12.5) | 52.7 (16.3) | 59.7 (8.8) | 59.3 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3 | 3 | 2 | 4 | 4 | 5 | 15 | 0 | 2 | 41
  Male | 2 | 2 | 4 | 6 | 2 | 2 | 9 | 3 | 0 | 3 | 4 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 5
  White | 3 | 3 | 6 | 8 | 3 | 5 | 12 | 6 | 14 | 3 | 5 | 68
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7 | 9 | 4 | 6 | 13 | 8 | 15 | 3 | 6 | 78

OUTCOME MEASURES:

1. Primary Outcome: Treatment-emergent Adverse Events (TEAEs) in Participants Regardless of Causality While Taking PLX3397 in Combination With Pembrolizumab
Description: Treatment-emergent Adverse Events (TEAEs) in participants regardless of causality while taking PLX3397 in combination with pembrolizumab are reported
Time Frame: 1 year (Dose Escalation); 2 years (Dose Expansion)
Population: Safety events were assessed in the Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: 400 mg/Day | Dose Escalation: 600 mg/Day | Dose Escalation: 600 mg/Day (Liver Metastases | Dose Escalation: 600 mg/Day (no Liver Metastases) | Dose Escalation: 800 mg/Day (Liver Metastases) | Dose Escalation: 800 mg/Day (no Liver Metastases) | Dose Expansion: Melanoma | Dose Expansion: NSCLC | Dose Expansion: Ovarian Cancer | Dose Expansion: SCCHN | Dose Expansion: GIST
Number analyzed (Participants) | 4 | 3 | 7 | 9 | 4 | 6 | 13 | 8 | 15 | 3 | 6
Participants | 4 | 3 | 7 | 9 | 4 | 6 | 12 | 8 | 15 | 3 | 6

2. Secondary Outcome: Summary of the Percentage of Participants With Objective Response Rate Assessed by RECIST v1.1 During Pembrolizumab and PLX3397
Description: Objective response rate was defined as the proportion of subjects who achieved a best disease response of either Complete or Partial (CR or PR) based on the Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed generally by MRI, CT, or PET-CT and are summarized as: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions. Participants who discontinued study therapy due to clinical progression, radiographic progression, or death without the required tumor assessments were considered to be non-responders in the Objective Response Rate (ORR) calculation. The efficacy analysis included all subjects with baseline tumor measurements who received at least 1 dose of study drug.
Time Frame: 1 year (Dose Escalation); 2 years (Dose Expansion)
Population: Overall best response was assessed in the Efficacy Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: 400 mg/Day | Dose Escalation: 600 mg/Day | Dose Escalation: 600 mg/Day (Liver Metastases | Dose Escalation: 600 mg/Day (no Liver Metastases) | Dose Escalation: 800 mg/Day (Liver Metastases) | Dose Escalation: 800 mg/Day (no Liver Metastases) | Dose Expansion: Melanoma | Dose Expansion: NSCLC | Dose Expansion: Ovarian Cancer | Dose Expansion: SCCHN | Dose Expansion: GIST
Number analyzed (Participants) | 4 | 3 | 7 | 9 | 4 | 6 | 13 | 8 | 15 | 3 | 6
Participants
  Complete response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial response | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0
  Progressive disease | 2 | 1 | 3 | 7 | 1 | 2 | 4 | 3 | 9 | 2 | 3
  Stable disease | 2 | 2 | 1 | 1 | 1 | 2 | 3 | 2 | 1 | 0 | 3
  Not evaluable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not assessed for response | 0 | 0 | 2 | 1 | 2 | 1 | 4 | 3 | 4 | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for each subject from after the first dose was administered to 30 days after the last dose, through study completion at Cycle 16 (up to approximately 100 weeks)
Description: Adverse events that emerge (or worsen) after the first dose of study drug and within 30 days after the last dose.
Arm/Group | Dose Escalation: 400 mg/Day | Dose Escalation: 600 mg/Day | Dose Escalation: 600 mg/Day (Liver Metastases | Dose Escalation: 600 mg/Day (no Liver Metastases) | Dose Escalation: 800 mg/Day (Liver Metastases) | Dose Escalation: 800 mg/Day (no Liver Metastases) | Dose Expansion: Melanoma | Dose Expansion: NSCLC | Dose Expansion: Ovarian Cancer | Dose Expansion: SCCHN | Dose Expansion: GIST
All-Cause Mortality (participants affected / at risk) | 2/4 | 2/3 | 2/7 | 6/9 | 2/4 | 0/6 | 5/13 | 1/8 | 3/15 | 1/3 | 0/6
Serious Adverse Events (participants affected / at risk) | 2/4 | 1/3 | 3/7 | 3/9 | 2/4 | 3/6 | 3/13 | 3/8 | 5/15 | 1/3 | 0/6
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 7/7 | 9/9 | 4/4 | 6/6 | 12/13 | 8/8 | 15/15 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation: 400 mg/Day (N=4) | Dose Escalation: 600 mg/Day (N=3) | Dose Escalation: 600 mg/Day (Liver Metastases (N=7) | Dose Escalation: 600 mg/Day (no Liver Metastases) (N=9) | Dose Escalation: 800 mg/Day (Liver Metastases) (N=4) | Dose Escalation: 800 mg/Day (no Liver Metastases) (N=6) | Dose Expansion: Melanoma (N=13) | Dose Expansion: NSCLC (N=8) | Dose Expansion: Ovarian Cancer (N=15) | Dose Expansion: SCCHN (N=3) | Dose Expansion: GIST (N=6)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Splenic infarction (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Obstruction gastric (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Parotitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radiation oesophagitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine with aura (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation: 400 mg/Day (N=4) | Dose Escalation: 600 mg/Day (N=3) | Dose Escalation: 600 mg/Day (Liver Metastases (N=7) | Dose Escalation: 600 mg/Day (no Liver Metastases) (N=9) | Dose Escalation: 800 mg/Day (Liver Metastases) (N=4) | Dose Escalation: 800 mg/Day (no Liver Metastases) (N=6) | Dose Expansion: Melanoma (N=13) | Dose Expansion: NSCLC (N=8) | Dose Expansion: Ovarian Cancer (N=15) | Dose Expansion: SCCHN (N=3) | Dose Expansion: GIST (N=6)
Anemia (All grades) (Blood and lymphatic system disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 5 | 1 | 6 | 2 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Leukopenia (All grades) (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Lymphadenopathy (All grades) (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Lymphopenia (All grades) (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (All grades) (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pancytopenia (All grades) (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Splenic infarction (All grades) (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (All grades) (Blood and lymphatic system disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Atrial fibrillation (All grades) (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Sinus bradycardia (All grades) (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Ear discomfort (All grades) (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Adrenal insufficiency (All grades) (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperthyroidism (All grades) (Endocrine disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (All grades) (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Uveitis (All grades) (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (All grades) (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (All grades) (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Abdominal pain (All grades) (Gastrointestinal disorders) | 1 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 5 | 1 | 2
Abdominal pain lower (All grades) (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 1 | 1 | 2 | 0 | 2 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breath odor (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chapped lips (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (All grades) (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 2 | 3 | 1 | 1
Defaecation urgency (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (All grades) (Gastrointestinal disorders) | 1 | 0 | 0 | 4 | 0 | 2 | 5 | 2 | 5 | 0 | 2
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry mouth (All grades) (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 0
Dysphagia (All grades) (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Faeces hard (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 0
Glossodynia (All grades) (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lower gastrointestinal hemorrhage (All grades) (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (All grades) (Gastrointestinal disorders) | 0 | 0 | 3 | 3 | 3 | 1 | 4 | 4 | 5 | 3 | 2
Obstruction gastric (All grades) (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Paraesthesia oral (All grades) (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (All grades) (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retching (All grades) (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Salivary gland enlargement (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Stomatitis (All grades) (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 1 | 0
Tongue discolouration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (All grades) (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1 | 2 | 3 | 5 | 3 | 1 | 1
Adverse drug reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 2 | 0
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (All grades) (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (All grades) (General disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 3 | 1 | 0 | 0 | 0
Decreased activity (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Device occlusion (All grades) (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Facial pain (All grades) (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (All grades) (General disorders) | 1 | 0 | 2 | 5 | 1 | 1 | 6 | 3 | 9 | 3 | 3
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Generalized oedema (All grades) (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza-like illness (All grades) (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malaise (All grades) (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Oedema peripheral (All grades) (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 0 | 0
Pain (All grades) (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 2 | 0 | 0
Peripheral swelling (All grades) (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Pyrexia (All grades) (General disorders) | 1 | 0 | 4 | 2 | 1 | 3 | 1 | 2 | 8 | 1 | 0
Bile duct obstruction (All grades) (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Drug-induced liver injury (All grades) (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic pain (All grades) (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperbilirubinemia (All grades) (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bacteremia (All grades) (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial infection (All grades) (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fungal infection (All grades) (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal skin infection (All grades) (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Furuncle (All grades) (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mastitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral candidiasis (All grades) (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Oral herpes (All grades) (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Parotitis (All grades) (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (All grades) (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rectal abscess (All grades) (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Root canal infection (All grades) (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Urinary tract infection (All grades) (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 2 | 0 | 0
Urinary tract infection bacterial (All grades) (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urosepsis (All grades) (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (All grades) (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (All grades) (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (All grades) (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion-related reaction (All grades) (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laceration (All grades) (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Procedure pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Radiation oesophagitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (All grades) (Investigations) | 0 | 2 | 1 | 1 | 1 | 3 | 5 | 3 | 9 | 1 | 4
Aspartate aminotransferase increased (All grades) (Investigations) | 1 | 2 | 2 | 4 | 2 | 3 | 6 | 3 | 8 | 1 | 4
Blood alkaline phosphatase increased (All grades) (Investigations) | 1 | 2 | 1 | 3 | 1 | 2 | 4 | 1 | 0 | 0 | 2
Blood bilirubin increased (All grades) (Investigations) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (All grades) (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 1
Blood creatinine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Blood potassium increased (All grades) (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (All grades) (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Breath sounds abnormal (All grades) (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Electrocardiogram PR prolongation (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram T wave abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (All grades) (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 1 | 3 | 0 | 1
Haemoglobin decreased (All grades) (Investigations) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Heart rate irregular (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Liver function test abnormal (All grades) (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mean cell haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mean cell volume decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neutrophil count decreased (All grades) (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 0
Nutritional condition abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Palpatory finding abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Platelet count decreased (All grades) (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0
Prothrombin time prolonged (All grades) (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thyroxine free decreased (All grades) (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Transaminase increased (All grades) (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0
Troponin increased (All grades) (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (All grades) (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 2 | 0
White blood cell count decreased (All grades) (Investigations) | 0 | 0 | 1 | 2 | 0 | 2 | 3 | 0 | 1 | 0 | 2
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (All grades) (Metabolism and nutrition disorders) | 1 | 0 | 3 | 3 | 1 | 2 | 4 | 3 | 6 | 1 | 1
Dehydration (All grades) (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 3 | 1 | 3 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (All grades) (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1 | 2 | 0 | 2 | 0 | 1 | 0 | 0
Hypomagnaesemia (All grades) (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Hyponatraemia (All grades) (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 2 | 2 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypophosphataemia (All grades) (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vitamin D deficiency (All grades) (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (All grades) (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 2 | 0 | 0
Back pain (All grades) (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 1 | 0 | 1 | 2 | 2 | 4 | 0 | 0
Flank pain (All grades) (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Groin pain (All grades) (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle oedema (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscular Stiffness (All Grades) (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscular weakness (All grades) (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (All grades) (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (All grades) (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 0
Myalgia (All grades) (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 1 | 2 | 0 | 0
Neck pain (All grades) (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 2 | 0 | 0 | 0
Pain in extremity (All grades) (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cancer pain (All grades) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (All grades) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Cerebral infarction (All grades) (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive disorder (All grades) (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (All grades) (Nervous system disorders) | 1 | 0 | 2 | 3 | 0 | 0 | 5 | 1 | 2 | 1 | 0
Dysarthria (All grades) (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (All grades) (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 1 | 1 | 0
Encephalopathy (All grades) (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage intracranial (All grades) (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (All grades) (Nervous system disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 3 | 2 | 1 | 1 | 0
Hydrocephalus (All grades) (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (All grades) (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine with aura (All grades) (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Paraesthesia (All grades) (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (All grades) (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (All grades) (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (All grades) (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Confusional state (All grades) (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hallucination (All grades) (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (All grades) (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Mental status changes (All grades) (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Haematuria (All grades) (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Proteinuria (All grades) (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urine abnormality (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Penile discharge (All grades) (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Perineal pain (All grades) (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alveolar lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (All grades) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0 | 3 | 4 | 5 | 5 | 1 | 0
Dysphonia (All grades) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Dyspnoea (All grades) (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 4 | 1 | 2 | 2 | 4 | 2 | 0 | 0
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea exertional (All grades) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 1 | 0
Epistaxis (All grades) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoptysis (All grades) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hypoxia (All grades) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal discharge discolouration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (All grades) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pharyngeal erythema (All grade) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (All grades) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 4 | 1 | 0
Pleuritic pain (All grades) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Pulmonary embolism (All grades) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhea (All grades) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Cold sweat (All grades) (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 1
Erythema (All grades) (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 0
Hair colour changes (All grades) (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0
Hyperhidrosis (All grades) (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Night sweats (All grades) (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (All grades) (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 3 | 5 | 0 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Rash (All grades) (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 3 | 1 | 0 | 0
Rash erythematous (All grades) (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash generalized (All grades) (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 0 | 1
Rash maculo-papular (All grades) (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 1 | 1 | 4 | 2 | 8 | 0 | 3
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Skin discolouration (All grades) (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin hyperpigmentation (All grades) (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin hypopigmentation (All grades) (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin lesion (All grades) (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 1 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (All grades) (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 2
Hypotension (All grades) (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Enrollment for this study was terminated early for insufficient evidence of clinical efficacy. Some of the planned statistical analyses described in the protocol and Statistical Analysis Plan (SAP) were not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/24/NCT02452424/Prot_SAP_000.pdf